CLINICAL TRIAL: NCT06237023
Title: The Impact of the Covid-19 Pandemic on Orthopedic Trauma Management; a Cross-sectional Study
Brief Title: The Impact of the Covid-19 Pandemic on Orthopedic Trauma Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Vedat Öztürk, MD, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 2021-168
Record Dates: First submitted 2024-01-30; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Trauma; COVID-19 Pandemic
MeSH Terms: conditions — Wounds and Injuries; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-pandemic group (Other): Patients who presented to the Orthopedics and Traumatology unit for any trauma-related reason during the one-year period prior to the pandemic
  Interventions: Other: epidemyolojical
- post-pandemic group (Other): Patients who presented to the Orthopedics and Traumatology unit for any trauma-related reason within one year from the start of the pandemic
  Interventions: Other: epidemyolojical

INTERVENTIONS:
Other: epidemyolojical — The aim of the study is to compare emergency orthopedic trauma admissions between the pre-pandemic and pandemic periods, and to identify changes in the epidemiology of orthopedic trauma.
  Other Names: Epidemiological

SUMMARY:
The aim of the study is to compare emergency orthopedic trauma admissions between the pre-pandemic period and the pandemic period and to detect changes in orthopedic trauma epidemiology.

DETAILED DESCRIPTION:
The aim of the study is to compare emergency orthopedic trauma admissions between the pre-pandemic period and the pandemic period and to detect changes in orthopedic trauma epidemiology. For this purpose, an epidemiological study was conducted in our country, comparing trauma admissions to a level 1 trauma hospital during a one-year period before the pandemic with those in the year following the onset of the pandemic.Demographic characteristics of the patients, such as age and gender, were recorded. In addition, the injury mechanisms of the patients, diagnosis, injured extremityor anatomical region, broken bone, fracture classification, multitrauma rates, trauma releated complications, hospitalization days, and treatment modalities were examined.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were admitted between March 2019 and March 2021
* Patients presenting due to trauma

Exclusion Criteria:

* Patients Admitted Before the Pandemic and Outside the Pandemic Period
* Consultation or Outpatient Clinic Patients
* Non-Traumatic Conditions
* Patients with Incomplete Records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57635 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Emergency Orthopedic Trauma Admissions Between Pre-Pandemic and Pandemic Period | up to 6 months
  The main purpose of the study is to compare the changes in the number and quality of emergency orthopedic trauma applications before the COVID-19 pandemic and during the pandemic period.
Detection of Changes in the Epidemiology of Orthopedic Trauma | up to 6 months
  The research aims to determine the changes in the epidemiology of orthopedic traumas during the pandemic period compared to before the pandemic. This includes patient demographics, injury mechanisms, diagnoses, injured extremity or anatomical sites, fracture types and classifications, polytrauma rates, trauma-related complications, length of hospital stay, and treatment methods.

SECONDARY OUTCOMES:
Changes in Patient Demographic Characteristics | 6 weeks
  Changes in the age and gender distribution of patients before the pandemic and during the pandemic period.
Comparison of Injury Mechanisms and Diagnoses | 8 weeks
  Different injury mechanisms and diagnosis distributions during the pandemic period compared to before the pandemic.
Injured Extremities or Anatomical Regions | 8 weeks
  The extremities or anatomical regions that were most frequently injured before and during the pandemic period.
Fracture Types and Classifications | 6 weeks
  Changes in fracture types and classifications during the pandemic period.
Trauma-Related Complications | 6 months
  Changes in trauma-related complication rates before the pandemic and during the pandemic period.
Treatment Methods | 8 weeks
  Changes in the treatment methods applied before the pandemic and during the pandemic period, especially the increases in surgical treatment rates.
Length of Hospital Stay | 6 weeks
  Differences in average length of hospital stay before the pandemic and during the pandemic period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Hamidiye Medical School, Bakırköy Dr. Sadi Konuk Education and Research Hospital, Department of Orthopedics and Traumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided